CLINICAL TRIAL: NCT03240796
Title: Secondary Intraocular Lens Implantation in Pediatric Patients: Minimal Invasive Surgery vs. Traditional Cataract Surgery for Treating Congenital Cataracts
Brief Title: Secondary Intraocular Lens Implantation in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPMOH2017-China-4
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Congenital Cataract
Keywords: congenital cataract; intra-capsular IOL implantation; ciliary sulcus fixation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimal invasive surgery and secondary IOL implantation (Experimental)
  Interventions: Procedure: minimal invasive surgery and secondary IOL implantation
- traditional cataract surgery and secondary IOL implantation (Active Comparator)
  Interventions: Procedure: traditional cataract surgery and secondary IOL implantation

INTERVENTIONS:
Procedure: minimal invasive surgery and secondary IOL implantation — We decreased the size of the capsulorhexis opening to 1.0-1.5 mm in diameter and moved the location of the capsulorhexis to the peripheral area of the lens instead of the central area. A 0.9 mm phacoemulsification probe was used to remove the lens contents and/or cortical opacities. Secondary IOL implantation: implant the IOL either into the capsule bag or fix at the ciliary sulcus.
  Arms: minimal invasive surgery and secondary IOL implantation
Procedure: traditional cataract surgery and secondary IOL implantation — traditional cataract surgery: anterior continuous capsulorhexis + irrigation/aspiration + posterior capsulorhexis + anterior vitrectomy (ACCC+ I/A + PCCC + Anti-vit).
  Secondary IOL implantation: implant the IOL either into the capsule bag or fix at the ciliary sulcus.
  Arms: traditional cataract surgery and secondary IOL implantation

SUMMARY:
This prospective, non-randomized controlled study aiming at comparing the prognosis of minimal invasive lens surgery and traditional cataract surgery for treating congenital cataracts after the patient receives secondary intraocular artificial lens (IOL) implantation.

DETAILED DESCRIPTION:
Pediatric patients received minimal invasive surgery and traditional lens removal surgery (anterior capsulorhexis and irrigation/aspiration and posterior capsulorhexis and anterior vitrectomy) are enrolled. The patients are assigned to two groups according to the strategy of primary surgery: Group I: the participants received minimal invasive surgery, while in Group II, the participants received a traditional cataract surgery. Investigators perform a secondary intraocular lens implantation for the patients. Investigators compare the visual acuity, incidence of high intraocular pressure, incidence of visual axis opacification, uveitis and iris/pupil abnormality between two groups after the first and the second surgery, aiming at comparing the prognosis of minimal invasive lens surgery and traditional cataract surgery for treating congenital cataracts.

ELIGIBILITY:
Inclusion Criteria:

Age between 24 months and 72 months Uncomplicated congenital cataract and underwent cataract removal Informed consent signed by a parent or legal guardian

Exclusion Criteria:

* Intraocular pressure >21 mmHg at enrollment Preterm birth (<28 weeks) Presence of other ocular diseases (keratitis, keratoleukoma, aniridia, glaucoma) or systemic disease (congenital heart disease, ischemic encephalopathy) History of ocular diseases (any congenital eye diseases, such as, congenital cataract, congenital glaucoma, congenital aniridia) in the family History of ocular trauma Microcornea Persistent hyperplastic primary vitreous Rubella Lowe syndrome

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | recorded at each follow-up (one week, one month, three months, six months after surgery, and every six months thereafter)
  measured using the Teller's acuity card, the Lea symbol visual acuity chart or the ETDRS chart according to the patient's age.

SECONDARY OUTCOMES:
Visual axis opacification | recorded at each follow-up (one week, one month, three months, six months after surgery, and every six months thereafter)
  Visual axis opacification was recorded by standardized slit lamp retroillumination.
High intraocular pressure | recorded at each follow-up (one week, one month, three months, six months after surgery, and every six months thereafter)
  measured with Tono-pen tonometer
Bi-ocular visual function | The examination is performed when the patient is four years old and older, once a year.
  determined with synoptophore

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D,Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center,Sun Yat-sen U, Guangzhou, Guangdong, China